CLINICAL TRIAL: NCT02023580
Title: Scale-up of an Internet-Delivered Randomized Controlled Trial for HIV+ Men
Brief Title: Scale-up of an Internet-Delivered Study for HIV+ Men
Acronym: Positive View
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Solutions (Other)
Collaborators: Hunter College of City University of New York (Other); Columbia University (Other); City University of New York, School of Public Health (Other); Emory University (Other)
Responsible Party: Principal Investigator, Sabina Hirshfield, Senior Research Scientist, Public Health Solutions
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH100973-01A1 (NIH)
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: HIV
Keywords: Viral suppression; Sexual risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The Video Treatment arm will complete baseline, 3-, 6-, 9-, and 12-month online survey assessments. Between baseline and 3-month follow-up, men will view 6 video vignettes (participants will receive a link to view a video vignette once a week for 6 weeks). Based on our team's experience of attenuated intervention effects at 6 months, men will receive 4 video boosters, spaced 1 week apart, after the 6-month assessment survey. Spacing the dose over time can improve critical thinking. The additional videos will be a continuation of the dramatic series plus additional video scenes on disclosure and serodiscordant partnerships.
  Interventions: Behavioral: Video treatments
- Control (Active Comparator): The video control arm will complete baseline, 3-, 6-, 9-, and 12-month online survey assessments. The control arm will receive the same number (and timing of) video clips as the intervention arm, but from a non-theoretically driven gay-oriented show with videos that are similar in length in order to preserve dosing equality across both arms. As the video treatment arm will be provided efficacious theory-driven videos, investigators expect to find a significant decrease in sexual risk behaviors in the intervention arm, compared to the control arm. Should this occur by month 6, with agreement from the data safety monitoring board (DSMB), investigators will provide the control arm with the video treatments.
  Interventions: Behavioral: Video treatments

INTERVENTIONS:
Behavioral: Video treatments — The treatment video vignettes to be delivered between Baseline and 3 Months include: 1) Condom use/anal sex without HIV status disclosure (potentially SDCAS); 2) Condom use/anal sex without HIV status disclosure and perceived responsibility; 3) Discussion of nondisclosure of HIV status prior to sex and perceived responsibility, STIs; 4) Stigma associated with disclosing HIV status to sex partners; 5) HIV/STI testing; and 6) Diagnosis of an STI; STI disclosure to sex partners and perceived responsibility.
  Video boosters to be delivered weekly for 4 weeks between 6 and 9 Months include: 7) HIV status disclosure, condom use, STIs; 8) STI disclosure to sex partners, disclosure to friends, serodiscordant partnerships; 9 & 10) Support of HIV disclosure and perceived responsibility.

SUMMARY:
Although HIV testing and highly effective antiretroviral therapy (ART) have improved survival with HIV, the relatively low level of ART adherence presents a significant public health challenge in terms of the potential to transmit HIV. Preventing transmission in virally unsuppressed HIV+ MSM who have condomless anal sex (CAS) with serodiscordant partners can have a great public health impact. As new HIV infections in MSM have been attributed in part to increased access to sex partners online, it is critical to deliver behavioral interventions to HIV+ MSM online to reach many high-risk men at a relatively low cost.

The investigators' theoretically-grounded HIV prevention videos about CAS, HIV disclosure, and testing in MSM were rigorously evaluated among MSM recruited online. Findings indicated significant reductions in CAS and significant increases in HIV status disclosure at 3-month follow-up, compared to baseline. In a subsequent online, randomized controlled trial (RCT) for MSM, investigators found significant reductions in CAS among MSM in the video arm at 60-day follow-up, compared to baseline; HIV+ MSM in the video arm reduced UAI, including serodiscordant CAS (SDCAS) at 60-day follow-up, compared to baseline. Based on these findings, investigators worked with POZ.com (POZ), the largest website for HIV+ individuals, to test whether they could recruit ethnically diverse HIV+ MSM and were very successful. The investigators have identified a potentially highly effective and feasible risk reduction intervention approach for HIV+ MSM.

With the commitment of POZ and a strong team of experts, the investigators propose to reshoot the videos to show the perspective of an HIV-positive man's experience with relationships and struggle ART adherence. The intervention videos will provide short doses for 10 online sessions (including boosters). We will target HIV+ MSM who are virally unsuppressed and monitor self-reported clinical indicators (i.e., viral load). Further, we will target online recruitment by race/ethnicity to enroll equal numbers of HIV+ White, Black and Hispanic MSM for balanced representation; improving retention with incentives and a proven online platform; including educational information about ART adherence; and cost and cost-effectiveness analyses for potentially averted HIV infections to determine health-related cost savings. Online, the investigators will recruit and follow a national sample of 1,500 high-risk, virally unsuppressed HIV+ MSM for 12 months.

DETAILED DESCRIPTION:
Study Design. For the primary outcomes (reduction in SDCAS and increase in HIV disclosure to sex partners), the proposed online study utilizes a 2-arm RCT design, with 10 intervention video vignettes grounded in SLT/SCT, to evaluate an innovative, multisession, video-based online intervention tailored to 1,500 English-speaking virally unsuppressed HIV+ White, Black and Hispanic MSM. Men will be randomized to receive 10 sessions of theory-driven video treatments or "attention" video controls. Men will be classified as White, Black, or Hispanic based on self-identification, and computerized randomization will occur within race/ethnicity to assure balanced representation across the experimental arms. All participants will receive online surveys at baseline, 3-, 6-, 9- and 12-month follow-up. All participants will receive incentives after completion of each online survey.

Preparation for Online RCT (AIM 1) (Months 1 - 12). In AIM 1 the investigators will finalize intervention materials for the RCT, plan online recruitment, program and test the online platform and work with the CAG to ensure appropriate literacy levels of the materials and surveys.

Theory-Driven Treatment Videos:

Employing a dramatic video series grounded in Social Learning and Social Cognitive theories, the Sex Positive![+] study engages learners through storytelling and promotes critical thinking on issues of HIV disclosure to sex partners, medication adherence and viral suppression, and serodiscordant condomless anal sex (CAS). In collaboration with a local production team, including a script writer, producer, and director, we produced Just a Guy, a six-episode video series that follows the story of "Guy", an openly gay man living with HIV in Brooklyn, NY. The video series is based, in part, on the HIV Big Deal project described above, which was launched online in 2008.

Attention Control Videos: The control arm receives ten healthy living videos that cover a range of topics including nutrition, physical exercise, smoking, and sleep quality. Attention control videos were selected from video-sharing websites and voted on by members of the research team.

Implementation of Online 2-Arm RCT (750/Arm) (AIM 2) (Months 17 - 35). In AIM 2 we will conduct the online 2-arm, video-based RCT, recruiting and randomizing 1,500 U.S. virally unsuppressed HIV+ White, Black and Hispanic MSM from POZ, Barebackrt, Facebook, Grindr and Craigslist. This 12-month online intervention has been designed to reduce high risk behavior using multi-session video vignettes and boosters.

Dissemination of the treatment and control videos will occur: 1) between baseline and 3-month follow-up, with men viewing 6 video vignettes, spaced 1 week apart; and 2) between 6- and 9-month follow-up, with men viewing 4 video boosters, spaced 1 week apart. *We will be able to track whether men click on the video links. All participants will complete baseline, 3-, 6-, 9-, and 12-month follow-up surveys. To reduce the chance of instrument reactivity (i.e., assessment effect), we will provide detailed online survey assessments at baseline and 12-month follow-up and brief online assessments at 3-, 6- and 9-month follow-up. All participants will receive a text or email with a link to the 3-, 6-, 9-, and 12-month follow-up surveys.

Arm 1: Video Treatment arm will complete baseline, 3-, 6-, 9-, and 12-month online survey assessments. Between baseline and 3-month follow-up, men will view 6 video vignettes (participants will receive a link to view a video vignette once a week for 6 weeks). Based on our team's experience of attenuated intervention effects at 6 months, men will receive 4 video boosters, spaced 1 week apart, after the 6-month assessment survey. Spacing the dose over time can improve critical thinking. The additional videos will be a continuation of the dramatic series plus additional video scenes on disclosure and serodiscordant partnerships.

Arm 2: Video Control arm will complete baseline, 3-, 6-, 9-, and 12-month online survey assessments. For comparability of study arms, the control group will be provided the same number of videos over the same time period.

The treatment video vignettes to be delivered weekly for 6 weeks between Baseline and 3 Months include: 1) Condom use/anal sex without HIV status disclosure (potentially SDUAI); 2) Condom use/anal sex without HIV status disclosure and perceived responsibility; 3) Discussion of nondisclosure of HIV status prior to sex and perceived responsibility, STIs; 4) Stigma associated with disclosing HIV status to sex partners; 5) HIV/STI testing; and 6) Diagnosis of an STI; STI disclosure to sex partners and perceived responsibility. Topics of the video boosters to be delivered weekly for 4 weeks between 6 and 9 Months include: 7) HIV status disclosure, condom use, STIs; 8) STI disclosure to sex partners, disclosure to friends, serodiscordant partnerships; 9 & 10) Support of HIV disclosure and perceived responsibility.

ART Adherence Content and Educational Messages. In response to the NIH review, we have expanded ART adherence-related content in the surveys for all participants (in addition to the adherence message they will see at the end of each survey). We will measure health literacy and numeracy, knowledge regarding clinical indicators, and self-efficacy to adhere to ART. A recent ART adherence study showed that, although low literate HIV+ patients were more likely to be non-adherent, self-efficacy mediated the impact of low literacy on ART adherence. We will conduct exploratory analyses of adherence with the social cognitive factors and primary outcomes.

Study Population. The target sample for this online RCT is 1,500 high-risk, virally unsuppressed HIV+ White, Black and Hispanic MSM in the US. Men will be identified via social networking (i.e., Facebook), sexual networking and dating websites (i.e., POZ.com, Barebackrt.com) as well as a GPS-based app (i.e., Grindr) and online classifieds (i.e., Craigslist). POZ is the largest site for HIV+ individuals and has 104,000 active MSM members. Barebackrt.com is the largest barebacking website for U.S. MSM with 56,305 unique monthly visitors. Grindr is the largest sexual networking GPS-based app with over 1.5 million U.S. users.

Inclusion Criteria. Subjects participating in any aspect of the study must report that they are 1) biologically male and identify their current gender as male; 2) age 18 or over; 3) able to read and respond in English; 4) reside within the U.S.; 5) report condomless anal sex with any HIV-negative or unknown status male partners in the past 6 months; 6) identify as HIV+; 7) in the past year, report a detectable viral load OR report not being on ART and not knowing their viral load OR report past month suboptimal ART adherence; 8) report their race and ethnicity as White, Black or Hispanic; 9) be willing to participate in an online intervention study for 12 months; and 10) have a working email address and cell phone number for intervention follow-up. We will employ quota sampling and targeted recruitment to ensure balanced representation of White (n=500), Black (n=500) and Hispanic (n=500) HIV+ MSM. Further, we will include the following Black racial/ethnic categories: Black, African American, Caribbean, African, or Multi-ethnic Black. Quota sampling and targeted recruitment will also be used to ensure representation of young MSM (18-29) in the sample (20%, n=300). All men enrolled in the study will be HIV+ by self-report, but health status will be less likely to influence participation since all study activities are online. Men who meet study criteria will automatically be randomized into 1 of the 2 study arms.

Exclusion Criteria. HIV-negative or untested MSM, women, transgendered persons, and anyone under age 18 will be excluded from the online study, as this is a study for biologically male virally unsuppressed HIV+ MSM; transgender women and biological females have different risk factors and sexual behaviors than MSM and deserve to have their own study. Further exclusions include those who are unwilling to provide key data (i.e., age, race and ethnicity, HIV status) on the online screener survey. Those who are found ineligible on the online screener survey will be informed that they are ineligible and thanked for their time. Those who drop out during the online screener, who refuse consent, or who drop out during online registration or before randomization will be considered non-responders. Those who drop out prior to completing the baseline assessment, but after study registration will be considered study applicants.

Online Recruitment (Months 17-23). As most online HIV prevention work has had low representation of minority MSM, we have set quotas to ensure balanced representation by race and ethnicity. To ensure recruitment goals are met for the racially/ethnically diverse U.S. sample of 1,500 virally unsuppressed HIV+ MSM, we will pursue multiple online venues for the online video-based RCT, which will also enable us to reach men with differing levels of connectedness to the HIV+ community. We will recruit equal numbers of HIV+ White (n=500), Black (n=500), and Hispanic (n=500) MSM.

* POZ.com recruitment. 104,000 POZ Personals members identify as gay (96,000) or bisexual (8,000) with the following racial/ethnic breakdown: 50% White (52,000), 20% Black (21,000), 12% Hispanic (12,000) and 18% mixed/other race (19,000). POZ.com will distribute e-mail blasts to POZ Personals members and will also recruit from their main webpage, Twitter account, and ads in their magazine.
* Facebook recruitment. We will simultaneously recruit on Facebook, as we may reach a different pool of HIV+ MSM on a social networking site. We have had success in recruiting racially/ethnically diverse HIV+ MSM from Facebook. For this study, we will use psychographic targeting (in-depth publicly available consumer data such as interests, occupation, and city).
* Bareback Real-Time Sex (Barebackrt.com). This U.S.-based hook-up site is for men seeking bareback sex (UAI). Barebackrt.com will work with us (sending emails to HIV+ members) at no cost.
* Craigslist. This free online classifieds service is one of the most popular websites in the U.S. and has been used successfully in our online work. For this study, research assistants will post ads on Craigslist in the Volunteers section and will repeatedly work his or her way through a targeted list of U.S. cities on Craigslist in order to reach a diverse (i.e., age, race and ethnicity) sample of MSM who reside outside of HIV epicenters.
* Grindr and Scruff. These GPS-based mobile (Smartphone) applications will target men in U.S. cities and towns to receive study advertisements (e.g., broadcast messages). Grindr will also distribute broadcast messages to users in Puerto Rico.
* BGCLive. Black Gay Chat is a sexual networking website with over 500,000 members. BGCLive will distribute e-mail blasts to its U.S. member base.
* MR X and Daddyhunt. We will purchase banner advertisements to appear online at Daddyhunt and on the mobile applications for MR X and Daddyhunt. We will also purchase broadcast messages to appear on the mobile applications for MR X and Daddyhunt.
* Wapo. We will purchase banner advertising to appear on the Wapo mobile application for gay and bisexual men. We will also purchase direct messaging to reach all U.S. users of the Wapo mobile application.
* Randomization. Once registration is completed, participants will automatically be randomized into 1 of 2 study arms. A computer program will assign each participant via stratified block randomization (by race/ethnicity and age) and will balance groups within a 5% range. Once men are randomized, they will begin the baseline survey. They be kept in their original assignment group (i.e., intent to treat) and be sent a link to the 3-, 6-, 9-, and 12-month follow-up surveys even if they do not participate in intervention activities. Randomization will be stratified by race/ethnicity and age (18-29, 30 and older), so that randomization will occur within each group (i.e., White, Black, or Hispanic). We will stop recruitment for HIV+ White MSM at 500, and over-sample HIV+ Hispanic MSM (n=500) and HIV+ Black MSM (n=500).

ELIGIBILITY:
Inclusion Criteria:

* biologically male
* age 18 or over
* able to read and respond in English
* reside within the U.S.
* report CAS with any HIV-negative or unknown status male partners in the past 6 months
* identify as HIV-positive
* in the past year, report a detectable viral load OR report not being on ART and not knowing their viral load OR report past month suboptimal ART adherence
* report their race and ethnicity as White, Black or Hispanic
* be willing to participate in an online intervention study for 12 months
* have a working email address and cell phone number for intervention follow-up

Exclusion Criteria:

* HIV-negative or untested MSM
* women
* transgender persons
* anyone under age 18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1197 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
SDCAS | 3 months, 6 months, 9 months, 12 months
  We will measure whether there is a reduction, increase, or no change in serodiscordant condomless anal sex with HIV-negative or unknown status male sex partners across the two study arms.

SECONDARY OUTCOMES:
HIV disclosure | 3 months, 6 months, 9 months, 12 months
  We will measure whether there is an increase, decrease or no change in HIV disclosure to sex partners across the two study arms at the above mentioned time frames.

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hirshfield, PhD, Principal Investigator — Public Health Solutions
Locations (1):
- Public Health Solutions, New York, New York, United States

REFERENCES:
- [Result] Yoon IS, Downing MJ Jr, Teran R, Chiasson MA, Houang ST, Parsons JT, Hirshfield S. Sexual risk taking and the HIV care continuum in an online sample of men who have sex with men. AIDS Care. 2018 Jul;30(7):921-929. doi: 10.1080/09540121.2017.1417535. Epub 2017 Dec 19. PMID 29258341
- [Result] Downing MJ Jr, Houang ST, Scheinmann R, Yoon IS, Chiasson MA, Hirshfield S. Engagement in Care, Psychological Distress, and Resilience are Associated with Sleep Quality among HIV-Positive Gay, Bisexual, and Other Men Who Have Sex with Men. Sleep Health. 2016 Dec;2(4):322-329. doi: 10.1016/j.sleh.2016.08.002. Epub 2016 Sep 19. PMID 28191491
- [Result] Hirshfield S, Downing MJ Jr, Parsons JT, Grov C, Gordon RJ, Houang ST, Scheinmann R, Sullivan PS, Yoon IS, Anderson I, Chiasson MA. Developing a Video-Based eHealth Intervention for HIV-Positive Gay, Bisexual, and Other Men Who Have Sex with Men: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2016 Jun 17;5(2):e125. doi: 10.2196/resprot.5554. PMID 27315764